CLINICAL TRIAL: NCT07169656
Title: Observation Study on Reducing the Risk of Liver Cancer Associated With Hepatitis B (Zhiyuan) Project.
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hongxia Liang, Chief physician, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: 2024-KY-0976-001
Record Dates: First submitted 2025-06-24; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: ETV,TDF,TAF,TMF
- Group 2
  Interventions: Drug: Peginterferon α-2b injection

INTERVENTIONS:
Drug: ETV,TDF,TAF,TMF — treated with entecavir (ETV), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide fumarate (TAF), or tenofovir amibufenamide (TMF)
  Groups: Group 1
Drug: Peginterferon α-2b injection — treated with Peginterferon α-2b injection
  Groups: Group 2

SUMMARY:
This study is a multicenter, prospective, observational real-world study designed to investigate and analyze the current treatment patterns of chronic hepatitis B (CHB) across 200 hospitals in China. By comparing patient outcomes under different therapeutic regimens, it aims to provide high-quality evidence-based medical data to optimize CHB treatment strategies and follow-up protocols, ultimately contributing to the advancement of a functional cure for chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* 1.Chronic HBV infection (HBsAg-positive for ≥6 months); 2.Age ≥18 years; 3.Patients who, based on real-world clinical practice needs, are planned or currently receiving treatment with:Entecavir (ETV),Tenofovir disoproxil fumarate (TDF),Tenofovir alafenamide fumarate (TAF),Tenofovir amibufenamide (TMF) OR Pegylated interferon α-2b-naïve patients OR Patients re-initiating pegylated interferon α-2b therapy; 4.Written informed consent obtained from the patient.

Exclusion Criteria:

* 1.Severe hepatic dysfunction or decompensated cirrhosis; 2.Concurrent participation in other clinical trials; 3.Hepatocellular carcinoma (HCC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were selected from chronic hepatitis B (CHB) cases across 200 national hospitals
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with HBsAg-associated HCC post-therapy | Week 4-240
Hepatocellular Carcinoma (HCC) Incidence | Week 4-240

SECONDARY OUTCOMES:
Number of chronic hepatitis B (CHB) patients with accurate knowledge/awareness of HBV | Week 4-240
Rate of HBsAg seroclearance | Week 4-240
HBsAg seroconversion rate | Week 4-240
Number of patients with altered HBsAg levels post-treatment | Week 4-240
Number of patients with HBsAg level decline from baseline | Week 4-240
HBeAg seroconversion rate | Week 4-240
HBV DNA | Week 4-240
Liver fibrosis improvement rate | Week 4-240
Incidence of liver cirrhosis | Week 4-240
Incidence of decompensated cirrhosis | Week 4-240
Incidence of decompensation-related complications | Week 4-240
Liver transplantation incidence rate | Week 4-240
Post-treatment relapse rate | Week 4-240

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Liang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (162):
- China (162):
  - Huaxian People's Hospital, Anyang
  - Linzhou City People's Hospital, Anyang
  - Neihuang County People's Hospital, Anyang
  - Tangyin County People's Hospital, Anyang
  - The Fifth People's Hospital of Anyang, Anyang
  - The First Affiliated Hospital of Xinxiang Medical University (Hua County Branch), Anyang
  - Guangzhou First People's Hospital, Guangzhou
  - The First Affiliated Hospital of Jinan University (Guangzhou Overseas Chinese Hospital), Guangzhou
  - Hebi Coal Mining Group General Hospital, Hebi
  - Hebi Infectious Disease Hospital, Hebi
  - Junxian County People's Hospital, Hebi
  - Bo'ai County People's Hospital, Jiaozuo
  - Mengzhou Hospital of Traditional Chinese Medicine, Jiaozuo
  - Qinyang People's Hospital, Jiaozuo
  - The Secend People's Hospital of Jiaozuo, Jiaozuo
  - The Third People's Hospital of Jiaozuo, Jiaozuo
  - Xiuwu People's Hospital, Jiaozuo
  - Wenxian People's Hospital, Jiayuguan
  - Jiyang County Hospital of Traditional Chinese Medicine, Jinan
  - Shandong Public Health Clinical Center, Jinan
  - Jiyuan People's Hospital, Jiyuan
  - Jiyuan Traditional Chinese Medicine Hospital, Jiyuan
  - Huaihe Hospital of Henan University, Kaifeng
  - Infectious Diseases Hospital of Kaifeng, Kaifeng
  - Kaifeng Central Hospital, Kaifeng
  - Kaifeng Hospital of Traditional Chinese Medicine, Kaifeng
  - Lankao First Hospital Group, Kaifeng
  - Qixian People's Hospital, Kaifeng
  - The People's Hospital of Weishi, Kaifeng
  - Tongxu County People's Hospital, Kaifeng
  - Weishi County People's Hospital, Kaifeng
  - Linyi Hospital of Traditional Chinese Medicine, Linyi
  - Linyi People's Hospital, Linyi
  - Linying County People's Hospital, Luohe
  - Luohe Central Hospital, Luohe
  - Luanchuan County People's Hospital, Luoyang
  - Luoning County People's Hospital, Luoyang
  - Luoyang Central Hospital, Luoyang
  - Luoyang First People's Hospital, Luoyang
  - Luoyang Third People's Hospital, Luoyang
  - Ruyang County People's Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Xin'an County People's Hospital, Luoyang
  - Yichuan County Hospital of Traditional Chinese Medicine, Luoyang
  - Yiyang County People's Hospital, Luoyang
  - Dengzhou Central Hospital, Nanyang
  - Dengzhou People's Hospital, Nanyang
  - Fangcheng County People's Hospital, Nanyang
  - Nanyang Central Hospital, Nanyang
  - Nanyang First People's Hospital, Nanyang
  - Nanyang Oilfield General Hospital, Nanyang
  - Nanyang Second General Hospital, Nanyang
  - Nanzhao County People's Hospital, Nanyang
  - Neixiang County People's Hospital, Nanyang
  - Sheqi County People's Hospital, Nanyang
  - Tanghe County People's Hospital, Nanyang
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Xinye County People's Hospital, Nanyang
  - Xixia County People's Hospital, Nanyang
  - Zhenping People's Hospital, Nanyang
  - Ningbo Medical Center Iihuili hospital, Ningbo
  - General Hospital Of Pingmei Shenma Group, Pingdingshan
  - Lushan County People's Hospital, Pingdingshan
  - People's Hospital of Baofeng, Pingdingshan
  - Pingdingshan First People's Hospital, Pingdingshan
  - Ruzhou First People's Hospital, Pingdingshan
  - Ye County People's Hospital, Pingdingshan
  - Pingdu Municipal People's Hospital, Pingdu
  - Anyang District Hospital, Pujiang
  - Chinese Medicine Hospital of puyang, Pujiang
  - Fanxian People's Hospital, Pujiang
  - Nanle County People's Hospital, Pujiang
  - Puyang People's Hospital, Pujiang
  - The Fifth People's Hospital of Puyang City, Pujiang
  - People's Hospital of Rizhao, Rizhao
  - Huanghe Sanmenxia Hospital, Sanmenxia
  - Sanmenxia Central Hospital, Sanmenxia
  - The First People's Hospital of Lingbao, Sanmenxia
  - The Sixth People's Hospital of Lingbao, Sanmenxia
  - Yimei Group General Hospital, Sanmenxia
  - Minquan County Hospital of Traditional Chinese Medicine, Shangqiu
  - Minquan County People's Hospital, Shangqiu
  - Second People's Hospital Xiayi Country, Shangqiu
  - Shangqiu Fourth People's Hospital, Shangqiu
  - Shangqiu Hospital of Traditional Chinese Medicine, Shangqiu
  - Shangqiu Municipal Hospital, Shangqiu
  - Shangqiu Third People's Hospital, Shangqiu
  - Sui County People's Hospital, Shangqiu
  - Suixian County Hospital of Traditional Chinese Medicine, Shangqiu
  - The First People's Hospital of Shangqiu, Shangqiu
  - The People's Hospital of Yucheng County, Shangqiu
  - Xiayi County People's Hospital, Shangqiu
  - Yongcheng Central Hospital, Shangqiu
  - Yucheng County People's Hospital, Shangqiu
  - Zhecheng People's Hospital, Shangqiu
  - Zhecheng Traditional Chinese Medicine Hospital Co., Ltd., Shangqiu
  - Changyuan County People's Hospital, Xinxiang
  - Huixian People's Hospital, Xinxiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Xinxiang First People's Hospital, Xinxiang
  - Xinxiang Infectious Disease Hospital, Xinxiang
  - Yanjin County People's Hospital, Xinxiang
  - Guangshan County People's Hospital, Xinyang
  - Gushi County People's Hospital, Xinyang
  - Huaibin County People's Hospital, Xinyang
  - Huangchuan County People's Hospital, Xinyang
  - Luoshan County People's Hospital, Xinyang
  - Xinyang Central Hospital, Xinyang
  - Xinyang Specialized Hospital for Infectious Diseases, Xinyang
  - Xixian People's Hospital, Xinyang
  - Changge People's Hospital, Xuchang
  - Xiangcheng County Traditional Chinese Medicine Hospital, Xuchang
  - Xiangcheng People's Hospital, Xuchang
  - Xuchang Central Hospital, Xuchang
  - Xuchang People's Hospital, Xuchang
  - Yanling County People's Hospital, Xuchang
  - Yanling County Traditional Chinese Medicine Hospital, Xuchang
  - Yuzhou Central Hospital, Xuchang
  - Yuzhou City People's Hospital, Xuchang
  - Chinese People's Liberation Army Joint Logistics Support Force 970 Hospital,, Yantai
  - Jiaozuo People's Hospital, Yantai
  - Yantai Qishan Hospital, Yantai
  - Gongyi City People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The First People's Hospit of Zhengzhou, Zhengzhou
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The Six People's Hospit of Zhengzhou, Zhengzhou
  - The Third People's Hospit of Zhengzhou, Zhengzhou
  - Third Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou
  - Xingyang People's Hospital, Zhengzhou
  - Zhengzhou Central Hospital, Zhengzhou
  - Zhengzhou Traditional Chinese Medicine Hospital, Zhengzhou
  - Zhongmu County Hospital of Traditional Chinese Medicine, Zhengzhou
  - Zhongmu County People's Hospital, Zhengzhou
  - Zhongshan Second People's Hospital, Zhongshan
  - Dancheng County People's Hospital, Zhoukou
  - Fugou County People's Hospital, Zhoukou
  - Shenqiu People's Hospital, Zhoukou
  - Taikang County People's Hospital, Zhoukou
  - The Frist People's Hospital Of Xiangcheng, Zhoukou
  - The People's Hospital Of Luyi, Zhoukou
  - Xihua County Hospital of Traditional Chinese Medicine, Zhoukou
  - Xihua County People's Hospital, Zhoukou
  - Zhoukou Central Hospital, Zhoukou
  - Zhoukou Hospital Of TCM, Zhoukou
  - Zhoukou Specialized Disease Hospital, Zhoukou
  - People's Hospital of Queshan, Zhumadian
  - Pingyu County People's Hospital, Zhumadian
  - Runan County Hospital of Traditional Chinese Medicine, Zhumadian
  - Shangcai County People's Hospital, Zhumadian
  - The 990th Hospital of the Joint Logistics Support Force of the PLA, Zhumadian
  - The People's Hospital Of Biyang Country, Zhumadian
  - Xincai County People's Hospital, Zhumadian
  - Xincai Medical University, Zhumadian
  - Xiping County People's Hospital, Zhumadian
  - Zhengyang County People's Hospital, Zhumadian
  - Zhumadian Central Hospital, Zhumadian
  - Zhumadian Traditional Chinese Medicine Hospital, Zhumadian
  - Zibo Central Hospital, Zibo
  - Zibo Infectious Diseases Hospital (Zibo Fourth People's Hospital), Zibo

IPD SHARING:
Plan to Share IPD: No